CLINICAL TRIAL: NCT00306189
Title: Dose Response Study of AMG 162 (Denosumab) in Subjects With Osteoporosis - A Randomized, Double-blind, Placebo-controlled, Dose Response Study of AMG 162 (Denosumab) in Japanese Postmenopausal Osteoporotic Subjects -
Brief Title: A Randomized, Double-blind, Placebo-controlled, Dose Response Study of AMG 162 (Denosumab) in Japanese Postmenopausal Osteoporotic Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20050172; NOT APPRICABLE
Record Dates: First submitted 2006-03-21; First posted 2006-03-23 (Estimated); Results first posted 2010-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Osteoporosis
Keywords: RANKL; RANK; denosumab; AMG 162; osteoporosis; bone turnover; bone mineral density; Japanese
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 100 mg AMG 162 (Active Comparator)
  Interventions: Drug: 100 mg AMG 162
- 60 mg AMG 162 (Active Comparator)
  Interventions: Drug: 60 mg AMG 162
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 14 mg AMG 162 (Active Comparator)
  Interventions: Drug: 14 mg AMG 162

INTERVENTIONS:
Drug: 100 mg AMG 162 — 100 mg AMG 162 (denosumab) SC every 6 months
  Arms: 100 mg AMG 162
Drug: 60 mg AMG 162 — 60 mg AMG 162 (denosumab) SC every 6 months
  Arms: 60 mg AMG 162
Drug: 14 mg AMG 162 — 14 mg AMG 162 (denosumab) SC every 6 months
  Arms: 14 mg AMG 162
Drug: Placebo — Placebo SC every 6 months
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the effect of AMG 162 (denosumab) treatment on the lumbar spine BMD at month 12 and safety profile across the dose range tested (14, 60 and 100 mg SC once every 6 months) in Japanese postmenopausal osteoporotic subjects compared with those treated with placebo over 12 months.

ELIGIBILITY:
Inclusion Criteria: - Ambulatory postmenopausal women. - BMD values (g/cm2, Hologic) must be lower than 0.714 at lumbar spine, 0.515 at femoral neck, 0.588 at total hip. - BMD values must not be lower than 0.535 at the lumbar spine, 0.406 at the femoral neck and 0.478 at the total hip. Exclusion Criteria: - Oral bisphosphonate treatments, PTH or PTH derivatives use within the last 12 months and administration of any of anti-osteoporotic treatments within the last 3 months before initial administration of the investigational product. - History of hypocalcemia. - More than two moderate vertebral fractures or any severe vertebral fracture.

Max Age: 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2006-01; Primary Completion 2007-06 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Nakamura T, Matsumoto T, Sugimoto T, Shiraki M. Dose-response study of denosumab on bone mineral density and bone turnover markers in Japanese postmenopausal women with osteoporosis. Osteoporos Int. 2012 Mar;23(3):1131-40. doi: 10.1007/s00198-011-1786-8. Epub 2011 Sep 17. PMID 21927920
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_49_AMG_162_20050172.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Placebo
Started | 57 | 56 | 56 | 57
Completed | 48 | 50 | 45 | 52
Not Completed | 9 | 6 | 11 | 5
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Adverse Event | 3 | 3 | 2 | 2
Not completed — Withdrawal by Subject | 4 | 2 | 8 | 1
Not completed — Ineligibility determined | 1 | 1 | 1 | 1
Not completed — Other | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Placebo | Total
Number analyzed (Participants) | 53 | 54 | 50 | 55 | 212
Age Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (7.1) | 65.1 (6.3) | 64.6 (7.1) | 64.6 (7) | 65.1 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 54 | 50 | 55 | 212
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Lumbar Spine Bone Mineral Density Percent Change From Baseline at Month 12
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 12 months
Population: All subjects who received >= 1 dose of investigational product and have a baseline and >= 1 post baseline measurement at the lumbar spine.
Measure: Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Placebo | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M
Number analyzed (Participants) | 55 | 53 | 54 | 50
Percent Change from Baseline | .46 [-.23 to 1.15] | 5.71 [4.76 to 6.65] | 6.73 [5.71 to 7.75] | 7.45 [6.38 to 8.53]
Statistical Analysis 1: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 7, 95% CI [5.76 to 8.24]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 5.25, 95% CI [4.1 to 6.4]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 6.27, 95% CI [5.06 to 7.49]

ADVERSE EVENTS:
Arm/Group | Placebo | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M
Serious Adverse Events (participants affected / at risk) | 4/54 | 6/53 | 4/54 | 2/51
Other Adverse Events (participants affected / at risk) | 49/54 | 50/53 | 47/54 | 48/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=54) | Denosumab 14 mg Q6M (N=53) | Denosumab 60 mg Q6M (N=54) | Denosumab 100 mg Q6M (N=51)
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebral artery embolism (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=54) | Denosumab 14 mg Q6M (N=53) | Denosumab 60 mg Q6M (N=54) | Denosumab 100 mg Q6M (N=51)
Palpitations (Cardiac disorders) | 0 | 0 | 3 | 1
Cataract (Eye disorders) | 1 | 3 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 5 | 5 | 2
Dental caries (Gastrointestinal disorders) | 4 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 2 | 3
Gastritis (Gastrointestinal disorders) | 0 | 1 | 3 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 1 | 3 | 1
Periodontitis (Gastrointestinal disorders) | 1 | 0 | 2 | 3
Stomach discomfort (Gastrointestinal disorders) | 3 | 3 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Malaise (General disorders) | 5 | 2 | 1 | 2
Seasonal allergy (Immune system disorders) | 3 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 3 | 0
Cystitis (Infections and infestations) | 3 | 2 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 3 | 1 | 2
Herpes zoster (Infections and infestations) | 1 | 4 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 21 | 18 | 22 | 22
Oral herpes (Infections and infestations) | 0 | 3 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 8 | 1 | 4 | 1
Joint sprain (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 5
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 8 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 6 | 1 | 1 | 1
Headache (Nervous system disorders) | 5 | 7 | 6 | 3
Hypoaesthesia (Nervous system disorders) | 3 | 1 | 2 | 5
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 3 | 6
Eczema (Skin and subcutaneous tissue disorders) | 5 | 6 | 4 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3
Hypertension (Vascular disorders) | 1 | 2 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.